CLINICAL TRIAL: NCT02844855
Title: Memory for Action in Neurological Patients
Acronym: EMBODIMENT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to recruit 83/99
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1608068; 2016-A00891-50 (Other: ANSM)
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease; Parkinson Disease
Keywords: Alzheimer; Parkinson; Action memory
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with Alzheimer disease (Active Comparator): Behavioral: Cognitive tests Only patients with Alzheimer disease will be included in this arm. Patients will perform different tasks : MMSE, (Folstein et al., 1975), HAD (Hospital Anxiety and Depression Scale; Zigmond & Snaith, 1983), a cognitive assessment (the 5 words test, Dubois et al., 2002; Trail Making test, Godefroy et al., 2008; BREF, Dubois et Pillon, 2000; Assessment of apraxia, Mahieux-Laurent, 2009) + the experimental task (verbal learning and action learning).
  Interventions: Behavioral: Cognitive tests
- patients with Parkinson disease (Active Comparator): Behavioral: Cognitive tests Only patients with Parkinson disease will be included in this arm. Patients will perform different tasks : MMSE, (Folstein et al., 1975), HAD (Hospital Anxiety and Depression Scale; Zigmond & Snaith, 1983), a cognitive assessment (the 5 words test, Dubois et al., 2002; Trail Making test, Godefroy et al., 2008; BREF, Dubois et Pillon, 2000; Assessment of apraxia, Mahieux-Laurent, 2009) + the experimental task (verbal learning and action learning).
  Interventions: Behavioral: Cognitive tests
- healthy controls (Sham Comparator): Behavioral: Cognitive tests Only patients with healthy controls will be included in this arm. Controls will perform different tasks : MMSE, (Folstein et al., 1975), HAD (Hospital Anxiety and Depression Scale; Zigmond & Snaith, 1983), a cognitive assessment (the 5 words test, Dubois et al., 2002; Trail Making test, Godefroy et al., 2008; BREF, Dubois et Pillon, 2000; Assessment of apraxia, Mahieux-Laurent, 2009) + the experimental task (verbal learning and action learning).
  Interventions: Behavioral: Cognitive tests

INTERVENTIONS:
Behavioral: Cognitive tests — MMSE, (Folstein et al., 1975), HAD (Hospital Anxiety and Depression Scale; Zigmond & Snaith, 1983), a cognitive assessment (the 5 words test, Dubois et al., 2002; Trail Making test, Godefroy et al., 2008; BREF, Dubois et Pillon, 2000; Assessment of apraxia, Mahieux-Laurent, 2009) + the experimental task (verbal learning and action learning).

SUMMARY:
Memory for action is especially important in everyday life although current literature is not very abundant. The enactment effect (i.e. better memory for performed actions than for verbally encoded sentences) is usually described as a robust effect in aging and can be found in many diseases. Although the enactment effect has been studied for three decades, there is still no consensus on how it enhances memory. Therefore, in order to gain additional insight into the representational basis of the enactment effect, in the present study, the investigators propose to test neurological patients. The investigators suggested that memory for action should be better than memory for verbally encoded information in Alzheimer's disease and Parkinson's disease.

If patients with Alzheimer's disease (AD) and Parkinson's disease (PD) have no cognitive assessment during the last 6 months, then they will realize different tests: MMSE (1), HAD (2), a cognitive assessment (3); (4); BREF (5); Assessment of apraxia, (6). Controls will perform the same tests to verify that they have no cognitive impairment. Then, two experimental conditions will be presented in all patients and controls: a first in which participants will have to name drawings (verbal learning) and a second in which they will have to reproduce an action associated with drawings (action learning). Immediately after this learning phase, a recognition task will be available and therefore participants will have to recognize drawings that had been presented previously. The main criteria used in the statistical analysis will be the correct recognition score.

DETAILED DESCRIPTION:
1. = Folstein et al., 1975,
2. = Zigmond & Snaith, 1983,
3. = Dubois et al., 2002;
4. = Godefroy et al., 2008;
5. = Dubois et Pillon, 2000;
6. = Mahieux-Laurent, 2009.

ELIGIBILITY:
Inclusion Criteria for 3 arms:

* Patient affiliated to a social security system
* Age between 55 and 80 years
* Normal vision and hearing or successfully corrected
* French mother tongue
* Signature of consent by participants

Specific criteria for inclusion of MA patients:

* Probable AD diagnosis made by a neurologist (McKhann et al., 2011)
* Mini-Mental State Examination (MMSE): score > 22
* Stable treatment for two months minimum.

Specific criteria for inclusion of PD patients:

* PD diagnosed by a neurologist (Postuma et al., 2015)
* Stable treatment for two months minimum.
* Mini-Mental State Examination (MMSE): score > 27
* Under dopaminergic treatment

Exclusion Criteria for 3 arms:

* Other neurological or psychiatric history
* Anxiety and depressive symptoms (assessed by the scale of depression-anxiety HAD; Zigmond & Snaith, 1983)
* Inability to communicate
* Significant impairment of judgment
* Delusional or psychotic state

Criteria common for non-inclusion of AD and PD patients:

* Other neurological or psychiatric history
* Anxiety and depressive symptoms (assessed by the scale of depression-anxiety HAD; Zigmond & Snaith, 1983)
* Inability to communicate
* Significant impairment of judgment
* Delusional or psychotic state

Criteria for non-inclusion of PD patients:

- Motor fluctuations

Criteria for non-inclusion of controls:

* Psychiatric or neurological disorders
* Anxiety and depressive symptoms (assessed by the scale of depression-anxiety HAD; Zigmond & Snaith, 1983)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-12-26 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Number of correct answers | Day 1
  The gain provided by the verbal learning vs action learning (number of correct answers).

CONTACTS AND LOCATIONS:
Overall Officials: Céline BORG, MD, Principal Investigator — celine.borg@univ-st-etienne.fr
Locations (2):
- France (2):
  - CHU de Saint-Etienne, Saint-Etienne
  - Hcl - Cm2R, Villeurbanne

IPD SHARING:
Plan to Share IPD: Undecided